CLINICAL TRIAL: NCT01528293
Title: A Prospective, Randomized, Comparative Effectiveness Trial of the ActiV.A.C.+ Compression Therapy Versus Compression Therapy Alone for the Treatment of Chronic Venous Ulcerations
Brief Title: ActiV.A.C.+ Compression Therapy Versus Compression Therapy Alone for the Treatment of Chronic Venous Ulcerations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment - unable to meet enrollment goals
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Christopher Attinger, M.D., Director, Wound Healing Clinic, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ActiVac
Record Dates: First submitted 2012-01-27; First posted 2012-02-08 (Estimated); Results first posted 2015-05-18 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Chronic Venous Hypertension With Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ActiVAC System+ Compression therapy (Active Comparator): ActiVAC System + Compression therapy group consisting of the application of this device along with compression therapy.
  Interventions: Device: ActiVAC System; Other: Compression therapy
- Compression therapy only (Other): Standard of Care compression therapy only
  Interventions: Other: Compression therapy

INTERVENTIONS:
Device: ActiVAC System — The ActiV.A.C. System will be applied in a customary manner per manufacturer's recommendations. Acticoat Flex 7™ will be applied as contact layer on the wound surface. Open cell foam is then applied over the top of the Acticoat Flex 7™. Adherent transparent occlusive material will be applied over the open cell foam. The tubing is then attached after cutting a small aperture through the occlusive material. Negative pressure will be set at 125mmHg on continuous suction. Sponge and canister will be replaced 2 time a week.
  Other Names: ActiV.A.C System
  Arms: ActiVAC System+ Compression therapy
Other: Compression therapy — Compression Therapy Profore™ multi-layered compression bandaging system will be utilized. This includes the application of a contact layer dressing using Acticoat Flex 7™. The compression bandage will be applied per manufacturer's recommendations.

SUMMARY:
This is a prospective, randomized, comparative interventional human subject trial. Patients with a chronic venous ulceration of the lower extremity will be enrolled into this study. These wounds must be recalcitrant to the standard treatment regimen. There are a total of two arms in this study. One group will be randomly assigned to receive Vacuum Assisted Closure (V.A.C. or VAC) by means of the ActiV.A.C. + Compression therapy group consisting of the application of this device along with compression therapy. The other group will be randomly assigned into compression therapy only group. A total of 60 subjects will be enrolled into this 6 week study. There will be a 2 week run-in period (prior to the onset of the intervention) to ensure that the wound has not healed greater than 35% prior to intervention and randomization. Wounds that heal within the 6 week trial period will have an additional confirmatory visit 2 weeks after healing was identified.

If within the 6 week intervention period the wound bed is determined to be ready for a Split Thickness Skin Graft (STSG) or Bio-engineered Alternative Tissue (BAT), the surgery or clinic application will be scheduled within 4 weeks. Subjects deemed not to be a surgical candidate, will have Bio-engineered Alternative Tissue (BAT) application in the clinic. This includes patients who are medically unstable to receive a medical clearance for surgery or otherwise not a candidate for Split Thickness Skin Graft (STSG) surgery (e.g. donor site skin is compromised). During this period between the scheduled STSG surgery or BAT application, the subjects will continue within the assigned treatment group. A confirmatory visit will also occur 2 weeks after the application of a Split Thickness Skin Graft (STSG) or Bio-engineered Alternative Tissue (BAT).

Patients diagnosed with a chronic venous ulceration will be assessed for study eligibility during their initial clinical evaluation. Patients who meet the eligibility requirements will be asked to enroll into the study (see Subject Recruitment). Subjects will be asked to sign the informed consent form and receive a copy of the informed consent.

DETAILED DESCRIPTION:
Patients diagnosed with a chronic venous ulceration will be assessed for study eligibility during their initial clinical evaluation. Patients who meet the eligibility requirements will be asked to enroll into the study (see Subject Recruitment). Subjects will be asked to sign the informed consent form and receive a copy of the informed consent. The study will be conducted in the following manner:

Prescreening, Screening, and Enrollment

* Obtain informed consent
* Assess patients for eligibility based on inclusion/exclusion criteria
* Initial quality of life questionnaire completed
* Target ulcer

  • If more than 1 wound is present on either leg; the target ulcer will be the one that is the largest in overall dimensions. All other ulcers will be treated per Standard of Care.
* Photo/wound measurements
* Venous studies (if necessary to confirm diagnosis)
* Case Record Form (CRF) completed
* Subjects will continue with Standard of Care until treatment initiation visit

  * If a patient is currently undergoing pump or pneumatic compression therapy, they must discontinue this treatment at least 2 week before the treatment initiation visit

Treatment Initiation Visit and Randomization

* Begin 2 weeks after the above enrollment visit - Confirm continued eligibility:

  * Photo/wound measurements (to be performed before and after debridement)
  * Exclude if wound size has decreased > 35% - Randomization into the 2 treatment groups

    1. ActiV.A.C. System Negative Pressure Therapy + Compression Therapy
    2. Compression Therapy - Quality of life questionnaires completed

       - CRF completed Subjects will have 1 visit in the clinic and 1 visit by a home nurse to change the dressing and Acti V.A.C ( if applicable) weekly

       Weekly Follow-Up
* Visits must be ± 2 days of scheduled appointment

  * Photo/wound measurements (to be performed before and after debridement)
  * Change ActiV.A.C. System+ Compression Therapy or Compression Therapy
  * Quality of life questionnaires to be completed at weeks 4, 6
  * CRF completed
  * If the subject is has not healed or healed, and the wound is not ready for a Split Thickness Skin Graft (STSG) or Bio-engineered Alternative Tissue (BAT)at the 6 week time point, then the patient will be exited from the study (see Close-Out)
  * If the subject has not healed within the 6 week interventional phase, but the wound is ready for a Split Thickness Skin Graft or Bio-engineered Alternative Tissue (BAT), they will be scheduled for a Split Thickness Skin Graft (STSG) or Bio-engineered Alternative Tissue (BAT)

Close-Out

* If the subject has not healed, they will be exited from the study at the 6 week time point
* Photo/wound measurements (to be performed before and after debridement)
* Close-out specific CRF completed
* Complete quality of life questionnaires
* Follow-up treatment plan with individual investigator

Confirmatory Visit

* If the target wound has healed within the 6 week interventional period, the subject will be scheduled for this confirmatory visit 2 weeks after wound has been deemed to be healed
* Photo/wound measurements (to be performed before and after debridement)
* Close-out specific CRF completed
* Complete quality of life questionnaires
* Follow-up treatment plan with individual investigator

Split Thickness Skin Graft (STSG) or Bio-engineered Alternative Tissue (BAT)- If the wound is deemed ready for Split Thickness Skin Graft (STSG) or Bio-engineered Alternative Tissue (BAT) then the subject will either:

* Be scheduled for surgery for application of a Split Thickness Skin Graft within 4 weeks
* Have Bio-engineered Alternative Tissue (BAT)applied in the clinic within 4 weeks

  * Subject will continue with their intervention until the date of surgery
  * After Split Thickness Skin Graft, subjects will receive Standard of Care (SOC) utilizing the ActiV.A.C. ™ + Compression Therapy
  * After Bio-engineered Alternative Tissue (BAT), subjects will receive Standard of Care utilizing compression therapy
  * Photo/Wound Measurements (to be performed before and after debridement)
  * CRF completed
  * Subjects will have a f/u visit within 5-7 days for dressing change per Standard of Care

Close-Out/Confirmatory Visit for Split Thickness Skin Graft (STSG) or Bio-engineered Alternative Tissue (BAT)

*2 weeks from the date of surgery (Split Thickness Skin Graft) or clinic application (Bio-engineered Alternative Tissue)

* Regardless if the target wound is healed or not, the subject will be exited from the study
* Photo/Wound measurements
* Percent adherence for subjects who received a Split Thickness Skin Graft
* Close-out specific CRF completed
* Complete quality of life questionnaires
* Follow-up treatment plan with individual investigator

Application of Devices/Dressing

The usual consent forms that are part of the Standard of Care will be utilized per the Center for Wound Healing at Georgetown University Hospital. All costs associated with the clinic visit consistent with the Standard of Care will be billed in the customary fashion.

Standard of Care Wound Therapy (Debridement, Infection Control)

The surface of the venous wound will be washed and rinsed with a wound cleanser at every visit per Standard of Care. The need for debridement (utilizing a scalpel and/or curette) will be dependent of the amount of nonviable tissue and/or biofilm detected on the surface of the wound. The decision to debride will be made by the individual investigator at each visit. The use of topical enzymatic debriding agents will be at the discretion of the investigator. Further, the investigator may use topical antimicrobials as needed. The use of oral antibiotics will also be at the discretion of the individual investigator. No other wound healing modalities including topically applied treatments will be allowed.

ActiV.A.C.® Therapy System

The ActiV.A.C.® Therapy System is an FDA approved device for the treatment of venous ulcerations. The ActiV.A.C.® System will be applied in a customary manner per manufacturer's recommendations. Acticoat Flex 7™ will be applied as the contact layer on the wound surface. Acticoat Flex 7™ is a fenestrated, silver-coated (anti-microbial), knitted polyester material that is routinely used as a contact layer dressing for chronic wounds. The open cell foam is then applied over the top of the Acticoat Flex 7™ (cut to shape of the wound). The adherent transparent occlusive material will be applied over the open cell foam. The tubing is then attached after cutting a small aperture through the occlusive material. Negative pressure will be set at 125 millimeters of mercury (mmHg) on continuous suction. The sponge and canister will be replaced 2 times per week. This dressing change will take place once in the clinic and once by the visiting home nurses. These nurses have had in-service training on the proper application of negative pressure therapy and have experience with its use.

Compression Therapy

Profore™ multi-layered compression bandaging system will be utilized. This includes the application of a contact layer dressing using Acticoat Flex 7™. The compression bandage will be applied per manufacturer's recommendations. The dressings will be changed 2 times per week. This dressing change will take place once in the clinic and once by the visiting home nurses. These nurses have had in-service training on the proper application of the compressive dressing and have experience with its use.

Standard of Care Post Split-Thickness Skin Graft or Application of a Bio-engineered Alternative Tissue (BAT)-

The application of a Split Thickness Skin Graft (STSG) or Bio-engineered Alternative Tissue (BAT) will follow the Standard of Care. This Standard of Care applies to both interventional groups. Split Thickness Skin Grafts will be applied in the operating room after debridement of the venous wound which will be conducted per Standard Of Care. After the placement of the Split Thickness Skin Graft onto the wound surface, a nonadherent dressing is placed onto the graft followed by a silver impregnated dressing layer. The ActiV.A.C.™ open celled foam will then be placed over the silver impregnated dressing in the customary fashion. Compressive dressing will then be placed over the ActiV.A.C.™ occlusive material. The postoperative dressings will be removed within 5-7 days. The wound site will then be redressed with a nonadherent dressing as the contact layer, silver impregnated dressing, and Profore™. The application of a BAT will take place in the outpatient clinic. This includes the debridement of the wound and the application of a Bio-engineered Alternative Tissue (BAT) onto the wound surface. The dressings include a nonadherent contact layer, followed by a silver impregnated dressing, and finally a Profore™ compressive dressing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 18-75 years of age
2. Subject able and willing to comply with study protocol requirements and able to understand the informed consent
3. Non-pregnant female willing to take urine pregnancy test
4. Chronic venous ulceration of the lower extremity

   * Defined: wound of greater than 1 month in duration
   * Diagnosis based on clinical assessment and/or venous studies
   * <100 cm2 area and <10cm at the widest diameter

Exclusion Criteria:

1. Active infection (redness, swelling, pain, purulence)
2. Untreated osteomyelitis or current osteomyelitis
3. Allergy or sensitivity to wound study products
4. Malignancy
5. Plantar surface wounds
6. BMI (Body Mass Index) ≥50
7. Uncontrolled diabetes (HbA1c>12%) at the time of study screening
8. End stage renal disease
9. Undergoing chemotherapy/radiation therapy
10. Non-dopplerable pedal pulses or otherwise diagnosed with peripheral arterial disease or any contraindication to compression therapy
11. Any previous wound care therapy including negative pressure therapy, ultrasound therapy, BAT, or STSG within the previous 30 days of enrollment; this excludes compression therapy
12. Greater than 35% wound surface area reduction in size at 2 weeks after initial screening visit
13. Pregnancy
14. Subject has any condition that, in the opinion of the investigator, makes the subject inappropriate to take part in this study
15. Subject unwilling or unable to comply with protocol requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Attinger, M.D, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, Center for Wound Healing, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ActiVAC System+ Compression Therapy: ActiVAC System + Compression therapy group consisting of the application of this device along with compression therapy.
  ActiVAC System + Compression therapy: The ActiV.A.C. System will be applied in a customary manner per manufacturer's recommendations. Acticoat Flex 7™ will be applied as contact layer on the wound surface. Open cell foam is then applied over the top of the Acticoat Flex 7™. Adherent transparent occlusive material will be applied over the open cell foam. The tubing is then attached after cutting a small aperture through the occlusive material. Negative pressure will be set at 125mmHg on continuous suction. Sponge and canister will be replaced 2 time a week.
  Compression Therapy Profore™ multi-layered compression bandaging system will be utilized. This includes the application of a contact layer dressing using Acticoat Flex 7™. The compression bandage will be applied per manufacturer's recommendations.
- Compression Therapy Only: Standard of Care compression therapy only
  ActiVAC System + Compression therapy: The ActiV.A.C. System will be applied in a customary manner per manufacturer's recommendations. Acticoat Flex 7™ will be applied as contact layer on the wound surface. Open cell foam is then applied over the top of the Acticoat Flex 7™. Adherent transparent occlusive material will be applied over the open cell foam. The tubing is then attached after cutting a small aperture through the occlusive material. Negative pressure will be set at 125mmHg on continuous suction. Sponge and canister will be replaced 2 time a week.
  Compression Therapy Profore™ multi-layered compression bandaging system will be utilized. This includes the application of a contact layer dressing using Acticoat Flex 7™. The compression bandage will be applied per manufacturer's recommendations.
Period: Overall Study
Arm/Group | ActiVAC System+ Compression Therapy | Compression Therapy Only
Started | 1 | 1
Completed | 0 | 1
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ActiVAC System+ Compression Therapy | Compression Therapy Only | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Compare Wound Healing
Description: Wound healing between the ActiV.A.C. System + Compression therapy versus Compression therapy alone in patients with chronic venous ulcerations.
Time Frame: 6 weeks
Population: Enrollment was insufficient to support statistical analyses. Three subjects were screened and only one completed the study.
Arm/Group | ActiVAC System+ Compression Therapy | Compression Therapy Only
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Compare the Time to Wound Bed Preparation, Quality of Life, Degree of Split Thickness Skin Graft/Bio-engineered Alternative Tissue Take
Description: -Compare the time to wound bed preparation between the ActiV.A.C. System + Compression therapy versus Compression therapy alone in patients with chronic venous ulcerations.
Time Frame: 9 weeks
Population: as for outcome 1
Arm/Group | ActiVAC System+ Compression Therapy | Compression Therapy Only
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: SF-12 Quality of Life Survey
Description: Quality of life between ActiV.A.C. System + Compression therapy versus Compression therapy alone in patients with chronic venous ulcerations.
Time Frame: 9 weeks
Population: as for outcome 1
Arm/Group | ActiVAC System+ Compression Therapy | Compression Therapy Only
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Degree of Take
Description: Degree of split thickness skin graft taken or bioengineered alternative tissue induced wound shrinkage after 6 weeks of ActiV.A.C. System + Compression therapy versus Compression therapy alone in patients with chronic venous ulcerations.
Time Frame: 6 Weeks
Population: as for outcome 1
Arm/Group | ActiVAC System+ Compression Therapy | Compression Therapy Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | ActiVAC System+ Compression Therapy | Compression Therapy Only
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Enrollment was insufficient to support statistical analyses. Three subjects were screened and only one completed the study. The study was terminated due to insufficient enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release but cannot embargo communications regarding trial results unless those communications are found inaccurate, contain Confidential Information, or would hinder seeking patent protection.